CLINICAL TRIAL: NCT05656911
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter Phase 2a Study to Investigate Efficacy and Safety of Zabedosertib (BAY 1834845) for the Treatment of Adult Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study to Learn How Well the Study Treatment Zabedosertib (BAY1834845) Works and How Safe it is Compared to Placebo in Adult Participants With Moderate-to-severe Atopic Dermatitis
Acronym: Damask
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22158; 2022-000520-38 (EudraCT Number)
Record Dates: First submitted 2022-11-29; First posted 2022-12-19 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — zabedosertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zabedosertib (Experimental): Participants will receive zabedosertib for up to 12 weeks (84 days).
  Interventions: Drug: Zabedosertib (BAY1834845)
- Matching placebo to zabedosertib (Placebo Comparator): Participants will receive placebo to zabedosertib for up to 12 weeks (84 days).
  Interventions: Drug: Placebo to zabedosertib (BAY1834845)

INTERVENTIONS:
Drug: Zabedosertib (BAY1834845) — Oral administration, two times a day
  Arms: Zabedosertib
Drug: Placebo to zabedosertib (BAY1834845) — Oral administration, two times a day
  Arms: Matching placebo to zabedosertib

SUMMARY:
Researchers are looking for a better way to treat atopic dermatitis (AD), an often long-lasting inflammation of the skin. Atopic dermatitis, also called eczema, is causing patches of skin to become swollen, red, cracked, and itchy.

The immune system helps protect the body from diseases. But sometimes the immune system can be too sensitive and overreact. This may then lead to allergies but also to skin conditions like atopic dermatitis.

The study treatment zabedosertib (BAY1834845) is currently under development for the treatment of atopic dermatitis and other inflammatory diseases. It works by reducing the activity of a protein called IRAK4. IRAK4 promotes the production and activation of a series of proteins that trigger inflammation reactions in the immune cells. By reducing the activity of IRAK4, the inflammation reactions are expected to be reduced.

The main purpose of the study is to learn how well zabedosertib works compared to placebo. A placebo is a treatment that looks like a medicine but does not have any medicine in it. How well it works means to find out the efficacy of zabedosertib. To answer this, the researchers will compare how many participants had 75% EASI score reduction after 12 weeks treatment between participants treated with zabedosertib and those treated with placebo. EASI represents Eczema Area and Severity Index (EASI). It is a tool for measuring the amount and severity of atopic dermatitis that a patient has on his or her body. The score ranges from 0-72, with 0 meaning clear skin and 72 meaning severe atopic dermatitis. In addition, the itch of the study participants and other tools for measuring the severity of atopic dermatitis will be assessed.

The secondary purpose of the study is to learn how safe it is compared to placebo. To know this, study team will compare how many participants having adverse events after taking study treatment between participants treated with zabedosertib and those treated with placebo.

In the study, participants will be randomly (by chance) assigned to receive zabedosertib or placebo. The participants from both treatment groups will take zabedosertib or placebo for up to 12 weeks.

The study consists of an up to 28-day screening period (Visits 1 and 2), a 12-week treatment period consisting of 5 visits (Visits 3 to 7), and a 4-week follow-up visits (Visits 8). Thus, the total study duration per participant will be 17 to 20 weeks (approximately 140 days).

During the study, the study team will:

* take blood and urine samples
* take skin samples (not obligatory for all patients)
* check the participants' disease area for assessment
* provide participants device to record their disease status and to take pictures on their disease areas
* have participants complete self-reported questionnaires
* do physical examinations
* examine heart health using ECG
* check vital signs
* ask the participants questions about how they are feeling and what events they are having.

An adverse event is any problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

At 28 days after the participants take their last treatment, the study team will check if participants have any events that might be related to the study treatment. This will be the last visit for the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of atopic dermatitis (AD) for ≥ 1 year at the screening visit.
* Moderate-to-severe AD at randomization visit as defined by

  * Eczema Area and Severity Index (EASI) score ≥ 16,
  * Body surface area (BSA) affected by AD ≥ 10%,
  * Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score ≥ 3, and
  * Peak Pruritus 0-10 numerical rating scale (NRS) ≥ 4 (average score of the daily scores of the 7 days before randomization, with ≥ 4 scores required).
* Documented history (within 6 months prior to the first screening visit) of inadequate response to treatment with topical corticosteroids (TCS), or if TCS are medically not advisable (e.g., due to important side effects or safety risks).
* Stable amount of emollient applied to skin over the whole body twice daily for at least the 7 consecutive days before the randomization visit
* Body mass index (BMI) within the range of 18.5 to 35.0 kg/m^2 (inclusive) at screening (Visit 1) and randomization visits.
* Women of childbearing potential and male subjects able to father children must agree to use adequate contraception when sexually active.

Exclusion Criteria:

* History of any major surgery within 8 weeks prior to screening or scheduled (elective) surgery, planned hospitalization and/or planned dental treatment during the study that could constitute a risk when participating in a study.
* Severe invasive infections in medical history and/or active clinically significant viral, bacterial, fungal, or parasitic infection (systemic or severe skin infection) ≤ 3 months prior to the randomization visit.
* A presence of uncontrolled condition including cardiovascular, respiratory, hepatic renal, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product, study conduct or could interfere with the interpretation of data.
* Known immunodeficiency disorder or immunocompromised state or, in the opinion of the investigator, unacceptable risk for participating in the study.
* Use of topical treatments for AD within 7 days before the randomization visit.
* Systemic immunosuppressive/ immunomodulating therapy or phototherapy within 4 weeks before the randomization visit.
* Therapy with biologic drugs within 5 half-lives of the biologic drug
* Known hypersensitivity to the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (4):
  - NorthShore University HealthSystem | Skokie Hospital - Dermatology Department, Skokie, Illinois
  - Beth Israel Deaconess Medical Center - Dermatology, Boston, Massachusetts
  - University of Cincinnati College of Medicine - Dermatology, Cincinnati, Ohio
  - Arlington Research Center, Inc. | Arlington, TX, Arlington, Texas
- Czechia (3):
  - Dermamedica s.r.o., Náchod, Královéhradecký kraj
  - Clintrial s.r.o., Prague
  - Praglandia, Prague
- France (3):
  - Clinique Bezannes, Bezannes
  - Centre Hospitalier Universitaire Nice | L'Archet Hospital - Dermatology Department, Nice
  - Hôpital Saint Louis, Paris
- Germany (2):
  - Hautarztpraxis Prof. Dr. med. Christian Termeer, Stuttgart, Baden-Wurttemberg
  - Charité - Universitätsmedizin Berlin, Berlin
- Italy (4):
  - A.O.U. di Ferrara, Ferrara, Emilia-Romagna
  - Humanitas Research Hospital | Cardio Center - Clinical, Interventional Cardiology and Coronary Care, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Policlinico G. Rodolico-San Marco Di Catania, Catania, Sicily
- Poland (4):
  - Dermal NZOZ Sp Osrodek Dermatologiczny Bialystok-Podlasie, Bialystok
  - Centrum Nowoczesnych Terapii Dobry Lekarz, Krakow
  - Santa Sp. z o.o., Lodz
  - Royalderm Agnieszka Nawrocka, Warsaw
- United Kingdom (2):
  - Whipps Cross University Hospital - Clinical Research Unit, Leytonstone, London
  - Medicines Evaluation Unit, Wythenshawe, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Jodl SJ, Worm M, Friedrichs F, Heinzel-Pleines U, Wagenfeld A, Feldmuller M, Klein S, Zhang R, Shakery K, Holzmann RD, Rohde B, Perera V. Efficacy and Safety of Zabedosertib, an Interleukin-1 Receptor-Associated Kinase 4 Inhibitor, in Patients with Moderate-to-Severe Atopic Dermatitis: A Phase II Randomized Study. Dermatol Ther (Heidelb). 2025 Nov;15(11):3329-3345. doi: 10.1007/s13555-025-01505-z. Epub 2025 Sep 4. PMID 40906353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 22 centers in Europe and US between 21-DEC-2022 (first participant first visit) and 31-JAN-2024 (last participant last visit).
Pre-assignment Details: A total of 129 participants were screened in this study. Of those, 52 did not pass screening (44 were screened failures, 1 was physician decision, 6 were subject decision, 1 was other reasons). A total of 77 participants were randomized.
Groups:
- Zabedosertib (BAY1834845): Participants received zabedosertib orally twice daily (BID) for 12 weeks (84 days).
- Placebo: Participants received matching placebo to zabedosertib orally twice daily (BID) for 12 weeks (84 days).
Period: Treatment Phase
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Started | 52 | 25
Completed | 36 | 19
Not Completed | 16 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 6 | 3
Not completed — Subject Decision | 4 | 2
Not completed — Other Reasons | 1 | 0
Not completed — Adverse Event | 3 | 1
Period: Follow-up Phase
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Started | 36 | 19
Completed | 35 | 18
Not Completed | 1 | 1
Not completed — Subject Decision | 0 | 1
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): All participants who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zabedosertib (BAY1834845) | Placebo | Total
Number analyzed (Participants) | 52 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (11.3) | 32.9 (10.3) | 34.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 7 | 33
  Male | 26 | 18 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 50 | 24 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 47 | 22 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Achievement of 75% Reduction From Baseline in the Eczema Area and Severity Index (EASI 75 Response) at Week 12 (Day 84)
Description: The endpoint was the composite variable defined as follows: - an EASI 75 response at Week 12 (Day 84), - no stop of study intervention for reasons related to lack of efficacy, - no rescue medication use during the 4 weeks before Day 84 and - no use of systemic atopic dermatitis (AD) treatment. The main estimand was the difference in the proportion of responders between treatment groups in adults with moderate-to-severe atopic dermatitis where use of topical rescue medication from Day 56 (Visit 6) onwards, use of systemic standard of care for AD and discontinuation of treatment due to lack of efficacy are handled as non-response (composite strategy). The estimand was regardless of use of rescue medication before Day 56 (Visit 6), regardless of non-compliance with emollients, and had treatment not been discontinued due to other reasons not related to lack of efficacy. Bayesian analysis according to estimand is presented.
Time Frame: Week 12 (Day 84)
Population: Per protocol set
Measure: Number; unit: Percentage (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Percentage (%) | 32.3 | 37.4
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; Median of posterior distribution of difference between Zabedosertib and Placebo including credible interval. Posterior probability is presented that the responder rate after treatment with zabedosertib is higher than after placebo given the data observed in the study; Test type: Other — Bayesian analysis according to estimand; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-29.0 to 18.0] — Posterior probability is 34.0%

2. Secondary Outcome: Percent Change From Baseline in EASI at Week 12 (Day 84)
Description: The EASI is a ClinRO assessing the extent of AD at four body regions by measuring the average severity of four clinical signs at each body region, each on a scale of 0 to 3. The minimum EASI score is 0 and the maximum EASI score is 72, with a higher score indicating worse severity of AD. The main estimand was based on the same strategies to address intercurrent events as described above for the primary endpoint. The mean difference between the treatment arms was used as summary measure.
Time Frame: Baseline and Week 12 (Day 84)
Population: Per protocol set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage (%) of change
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
percentage (%) of change | -44.58 [-55.96 to -33.19] | -55.88 [-71.91 to -39.85]
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; The analysis of covariance (ANCOVA) model includes treatment group as fixed effect and the EASI baseline value as covariate; Test type: Other; p = 0.257, ANCOVA — two-sided. No adjustment for multiple comparisons; Mean Difference (Final Values) = 11.31, 95% CI 2-sided [-8.26 to 30.87] — LS mean (%)

3. Secondary Outcome: Achievement of EASI 50 Response at Week 12 (Day 84)
Description: The EASI is a ClinRO assessing the extent of AD at four body regions by measuring the average severity of four clinical signs at each body region, each on a scale of 0 to 3. The minimum EASI score is 0 and the maximum EASI score is 72, with a higher score indicating worse severity of AD. EASI 50 corresponds to the achievement of 50% reduction from baseline in EASI. The main estimand was calculated similarly as for EASI 75. Bayesian analysis according to estimand is presented.
Time Frame: Week 12 (Day 84)
Population: Per protocol set
Measure: Number; unit: Percentage (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Percentage (%) | 52.7 | 55.4
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Bayesian analysis according to estimand; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-27.0 to 22.1] — Posterior probability is 41.7%

4. Secondary Outcome: Achievement of EASI 90 Response at Week 12 (Day 84)
Description: The EASI is a ClinRO assessing the extent of AD at four body regions by measuring the average severity of four clinical signs at each body region, each on a scale of 0 to 3. The minimum EASI score is 0 and the maximum EASI score is 72, with a higher score indicating worse severity of AD. EASI 90 corresponds to the achievement of 90% reduction from baseline in EASI. The main estimand was calculated similarly as for EASI 75. Bayesian analysis according to estimand is presented.
Time Frame: Week 12 (Day 84)
Population: Per protocol set
Measure: Number; unit: Percentage (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Percentage (%) | 15.6 | 20.4
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Bayesian analysis according to estimand; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-25.6 to 13.4] — Posterior probability is 31.5%

5. Secondary Outcome: Achievement of a vIGA-AD Response (Score 0 or 1 and ≥ 2 Points Improvement) at Week 12 (Day 84)
Description: vIGA-AD stands for validated Investigator Global Assessment for Atopic Dermatitis. The vIGA-AD is a 1-item static ClinRO using a 5-point scale from 0 (clear) to 4 (severe) based on 4 clinical features of AD lesions: erythema, induration/papulation, lichenification, and oozing/crusting, and takes extent of disease into account. The main estimand was calculated similarly as for EASI 75. Bayesian analysis according to estimand is presented.
Time Frame: Week 12 (Day 84)
Population: Per protocol set
Measure: Number; unit: Percentage (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Percentage (%) | 15.9 | 28.5
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Bayesian analysis according to estimand; Mean Difference (Final Values) = -12.5, 95% CI 2-sided [-34.1 to 7.0] — Posterior probability is 10.8%

6. Secondary Outcome: Absolute Change From Baseline in Body Surface Area (BSA) Affected by Atopic Dermatitis (AD) at Week 12 (Day 84)
Description: BSA affected by AD was assessed for each section of the body, e.g. using the rule of nines. The possible highest score for each region is: Head and neck - 9%; Anterior trunk - 18%; Back - 18%; Upper limbs - 18%; Lower limbs - 36%; Genitals - 1%. Affected BSA was reported as a percentage of all major body sections combined. The main estimand was based on the same strategies to address intercurrent events as described above for the primary endpoint. The mean difference between the treatment arms was used as summary measure.
Time Frame: Baseline and Week 12 (Day 84)
Population: Per protocol set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of BSA (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
percentage of BSA (%) | -13.28 [-18.98 to -7.58] | -20.34 [-28.60 to -12.07]
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.166, ANCOVA — two-sided. No adjustment for multiple comparisons; Mean Difference (Final Values) = 7.06, 95% CI 2-sided [-2.92 to 17.03]

7. Secondary Outcome: Achievement of a ≥ 4 Point-improvement (Reduction) in the Weekly Average of the Peak Pruritus 0-10 NRS Score From Baseline to Week 12 (Day 84) for Participants With Peak Pruritus 0-10 NRS Score ≥ 4 at Baseline
Description: NRS stands for numerical rating scale. The Peak Pruritus 0-10 NRS is a single patient-reported item designed to measure peak pruritus (itch), or 'worst' itch, over the previous 24 h based on the following question: 'On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable", how would you rate your itch at the worst moment during the previous 24 hours?'. ≥ 4 points reduction of the Peak Pruritus 0-10 NRS is considered a clinically relevant within-person response. NRS was assessed on a daily basis and the average over the last 7 days before the visit day was used for analysis. The main estimand was calculated similarly as for EASI 75. Bayesian analysis according to estimand is presented.
Time Frame: Baseline and Week 12 (Day 84)
Population: Per protocol set
Measure: Number; unit: Percentage (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Percentage (%) | 16.4 | 25.0
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Bayesian analysis according to estimand; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-30.4 to 11.0] — Posterior probability is 20.5%

8. Secondary Outcome: Absolute Values of Weekly Average of the Peak Pruritus 0-10 Numerical Rating Scale (NRS) Score at Week 12 (Day 84)
Description: The Peak Pruritus 0-10 NRS is a single patient-reported item designed to measure peak pruritus (itch), or 'worst' itch, over the previous 24 h based on the following question: 'On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable", how would you rate your itch at the worst moment during the previous 24 hours?'. ≥ 4 points reduction of the Peak Pruritus 0-10 NRS is considered a clinically relevant within-person response. NRS was assessed on a daily basis and the average over the last 7 days before the visit day was used for analysis. The main estimand was based on the same strategies to address intercurrent events as described above for the primary endpoint.
Time Frame: Week 12 (Day 84)
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
Scores on a scale | 5.759 (2.218) | 5.36 (2.311)

9. Secondary Outcome: Percent Change of Weekly Average of the Peak Pruritus 0-10 NRS Score From Baseline at Week 12 (Day 84)
Description: The Peak Pruritus 0-10 NRS is a single patient-reported item designed to measure peak pruritus (itch), or 'worst' itch, over the previous 24 h based on the following question: 'On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable", how would you rate your itch at the worst moment during the previous 24 hours?'. ≥ 4 points reduction of the Peak Pruritus 0-10 NRS is considered a clinically relevant within-person response. NRS was assessed on a daily basis and the average over the last 7 days before the visit day was used for analysis. The main estimand was based on the same strategies to address intercurrent events as described above for the primary endpoint. ANCOVA analysis according to estimand is presented.
Time Frame: Baseline and Week 12 (Day 84)
Population: Per protocol set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change (%)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 47 | 22
percentage of change (%) | -20.65 [-29.54 to -11.77] | -27.33 [-40.00 to -14.66]
Statistical Analysis 1: Comparison: Zabedosertib (BAY1834845) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.396, ANCOVA — two-sided. No adjustment for multiple comparisons; Mean Difference (Final Values) = 6.68, 95% CI 2-sided [-8.75 to 22.11]

10. Secondary Outcome: Frequency and Severity of Treatment-emergent Adverse Events (TEAEs)
Time Frame: From first treatment with the study intervention until 7 days after the last intake of study intervention (approximately up to 91 days)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Zabedosertib (BAY1834845) | Placebo
Number analyzed (Participants) | 52 | 25
Participants
  Any AE | 23 | 7
  Maximum intensity for any AE -MILD | 13 | 4
  Maximum intensity for any AE -MODERATE | 10 | 3
  Any SAE | 0 | 0
  AE with outcome death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events tables: from the start of study intervention until 7 days after the last intake (approximately up to 91 days). All-cause mortality is considered after signing informed consent up to the last contact per participant, up to 20 weeks.
Groups:
- Zabedosertib (BAY1834845): Participants received zabedosertib for up to 12 weeks (84 days)
- Placebo: Participants received matching placebo to zabedosertib for up to 12 weeks (84 days)
Arm/Group | Zabedosertib (BAY1834845) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/25
Other Adverse Events (participants affected / at risk) | 23/52 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zabedosertib (BAY1834845) (N=52) | Placebo (N=25)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Pustule (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Eczema impetiginous (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pregnancy of partner (Social circumstances) | 0 (0) | 1 (1)
Gingival graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings by the sponsor. If this is foreseen by the investigator, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT05656911/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT05656911/SAP_001.pdf